CLINICAL TRIAL: NCT02444312
Title: A Randomised Controlled Trial of Benefit Finding in Caregivers: The Building Resources in Caregivers (BRiC) Study Protocol
Brief Title: Trial of Benefit Finding in Caregivers: The Building Resources in Caregivers (BRiC) Study
Acronym: BRiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Carolan Research Institute (Unknown); Care Alliance Ireland (Unknown)
Responsible Party: Principal Investigator, Brenda O'Connell, Ms. Brenda O'Connell, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRiC2015
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Quality of Life; Psychological Distress
Keywords: Caregiving; Benefit Finding; Writing Intervention

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benefit-finding Writing Activity (Experimental): For two weeks, on six days of their choice, caregivers will be instructed to write about their thoughts and feelings in a diary/ notebook about the benefits of caring.
  Interventions: Behavioral: Benefit-finding Writing Activity
- Neutral Writing activity (Active Comparator): For two weeks, on six days of their choice, caregivers will be instructed to write about a neutral topic.
  Interventions: Behavioral: Neutral Writing Activity

INTERVENTIONS:
Behavioral: Benefit-finding Writing Activity — Caregivers will be instructed to write about the benefits of caring, considering things such as improved social relationship, appreciation of life and loved ones, and the positive consequences with respect to these.
  Arms: Benefit-finding Writing Activity
Behavioral: Neutral Writing Activity — The control group will be instructed to write number of things about the weather that day. Although the sentences can be as long or as short as they like, they will be encouraged to try and aim for about 3 or 4 sentences at least.
  Arms: Neutral Writing activity

SUMMARY:
A randomised controlled trial that will compare the effects of a brief benefit -finding writing intervention with an active control condition on quality of life and psychological health among informal caregivers.

DETAILED DESCRIPTION:
A double-blind, randomized controlled parallel group study design with an equal 1:1 allocation ratio will be employed. This study will compare the effect of a brief benefit finding writing intervention with a control condition among caregivers. Caregivers currently caring for people with mental and physical disabilities will be randomised into a two-week, a) a benefit writing group or b) a control writing group. Caregivers will complete self-report measures relating to their care-recipient and themselves (e.g., illness type, and sociodemographics) and psychometric measures of benefit finding (primary outcome), psychological distress and quality of life(secondary outcomes). These will be assessed via online software at baseline, immediate post-test and at 3 month follow-up. Additionally, expectations and fidelity indices will be assessed and qualitative commentary on participation experiences gathered.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 18
* Must identify as caring for a family member, friend or relative
* Must be living in Ireland

Exclusion Criteria:

* If the person cared for is living in institutional care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Benefit Finding (Adapted version of the 17-item Benefit Finding Scale; Antoni et al., 2001) | Baseline, immediate post-intervention (two weeks), and 3 months
  Used to assess change in benefit-finding levels over the course of the intervention and follow-up

SECONDARY OUTCOMES:
Caregiver Quality of Life (40 item Adult Carer Quality of Life Questionnaire; Joseph, Becker, Elwick, & Silburn, 2012) | Baseline, immediate post-intervention (two weeks), and 3 months
  This measures quality of life in eight separate domains: support for caring; caring choice; caring stress; money matters; personal growth; sense of value; ability to care; and carer satisfaction. Used to assess change in quality of life levels over the course of the intervention and follow-up
Psychological Distress (Hospital and Anxiety Depression Scale; Zigmond & Snaith, 1983) | Baseline, immediate post-intervention (two weeks), and 3 months
  Used to assess change in psychological distress levels over the course of the intervention and follow-up, and as a moderator

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gallagher, PhD, Study Director — University of Limerick, Department of Psychology; Charles Brand, MSc, Principal Investigator — University of Limerick; Brenda H O' Connell, B.A, Principal Investigator — University of Limerick